CLINICAL TRIAL: NCT03557658
Title: A Phase 1, Open-label, Parallel-group Study to Evaluate the Effect of Moderate Hepatic Impairment on the Pharmacokinetics and Pharmacodynamics of Bexagliflozin
Brief Title: Safety and Efficacy of Bexagliflozin in Subjects With Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THR-1442-C-455
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — bexagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hepatic Impaired (Experimental): Subjects with hepatic impairment conforming to the Child-Pugh class B (total score 7-9)
  Interventions: Drug: Bexagliflozin
- Healthy Volunteer (Experimental): Subjects with normal hepatic function
  Interventions: Drug: Bexagliflozin

INTERVENTIONS:
Drug: Bexagliflozin — Single oral dose of bexagliflozin tablet, 20 mg

SUMMARY:
The purpose of this study is to examine the drug exposure and drug effects on subjects with moderate hepatic impairment after a single oral dose of bexagliflozin tablets, 20mg. The study will also evaluate how safe the study drug is and how well the study drug is tolerated in subjects with moderate hepatic impairment.

DETAILED DESCRIPTION:
This was a Phase 1, open-label, parallel-group study designed to assess the effect of moderate hepatic impairment on the PK and PD of orally administered bexagliflozin tablets. A total of 16 subjects comprising eight with moderate hepatic impairment (Child Pugh total score 7 to 9) and eight healthy, matched controls, were enrolled and received a single oral dose of bexagliflozin tablets, 20 mg, after an overnight fast. Food was withheld for at least 2 h after dosing. Water was allowed as desired except within 1 h of drug administration.

Blood samples were collected prior to dosing, and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h post-dose.

The unbound fraction of bexagliflozin at 24 h post dose and at the maximum plasma concentration for each subject was determined by equilibrium dialysis.

Urine samples for PD analysis were collected for the 12 h interval preceding dosing and for the 0 - 12 h, 12 - 24 h, 24 - 36 h, and 36 - 48 h intervals following dosing.

ELIGIBILITY:
Each subject had to meet the following criteria to be eligible for the study:

1. Be male or female adults between the age of 18 and 75 years
2. Have a body mass index (BMI) of 18.0 kg/m2 to 40.0 kg/m2
3. Have adequate venous access at multiple sites in both arms
4. Be willing to be confined to the clinical research facility as required by the protocol
5. Be able to comprehend the explanation of the informed consent and be willing to provide written informed consent in accordance with institutional and regulatory guidelines
6. For subjects in the hepatic impairment group only: Be diagnosed with moderate hepatic impairment with a Child-Pugh score 7 to 9 and be in stable general health apart from hepatic impairment and its related conditions.
7. For subjects in the healthy control group only:

   * Be in general good health with matching demographics and baseline characteristics to individual subjects in the hepatic impairment group by age (± 10 years), weight (± 10%), sex, and smoking status
   * Exhibit neither evidence of an active infection nor undergoing any treatment with antibiotics at the time of Screening.

Prospective subjects who met any of the following criteria were ineligible to participate:

1. A clinically significant history of allergy to drugs or latex
2. A positive alcohol or drug result based on urine sample or breathalyzer testing at Screening or at clinic admission
3. A donation of 400 mL of whole blood within two months, 200 mL of whole blood within one month, or blood components or plasma within 14 days prior to Day 0
4. A history of exposure to an investigational drug within 30 days or 5 half-lives of the investigational drug prior to Day 0, whichever was longer
5. A history of exposure to any SGLT2 inhibitor within 3 months prior to Day 0 or participation in previous bexagliflozin clinical trials
6. A history of exposure to probenecid, rifampin, or any potential strong UGT1A9 inducers or inhibitors within 2 months of Day 0
7. A clinically significant abnormal electrocardiogram (ECG) that includes but is not limited to: heart rate < 40 or > 110 bpm, QRS> 160 ms, QTc> 480 ms (corrected by Bazett's formula), or any clinically significant arrhythmia including Mobitz type II 2nd Degree Heart block and bifascicular block
8. A history of human immunodeficiency virus (HIV) infection or a positive titer for HIV antibody
9. A history of vaccination (with the exception of the flu vaccine) within 30 days prior to Day 0
10. An estimated glomerular filtration rate (eGFR) < 60 mL·min-1 per 1.73 m2 as calculated by the modification of diet in renal disease study equation
11. Severe or moderate renal dysfunction or a history of kidney, other organ, bone marrow, or stem cell transplant
12. If male, unwilling to refrain from donating sperm or to use appropriate birth control when engaging in sexual intercourse for the duration of the study and a period of 14 days after discharge from the clinic. Surgically sterile male subjects were eligible
13. If female and of childbearing potential, unwilling to use an adequate method of contraception to avoid or prevent pregnancy for the duration of the study and 14 days after discharge from the clinic. Surgically sterile (as a result of hysterectomy or bilateral oophorectomy), or postmenopausal (absence of menses greater than 12 months and age > 45 years) female subjects were eligible. All females were to have had a negative pregnancy test at Screening and at clinic admission
14. Unwillingness to forgo consumption of grapefruit and grapefruit products from 7 days prior to Day 0 through discharge from the clinic
15. Pre existing thrombocytopenia (platelet blood count < 30,000 platelets) at Screening or other clinically significant findings in complete blood count (CBC) test.
16. A history of current febrile illness, hepatocellular carcinoma, acute liver disease, severe hepatic encephalopathy, or biliary liver cirrhosis.
17. A history of significant acute medical illness (new conditions and/or exacerbation of pre existing conditions or major surgery within 4 weeks of study drug administration), active alcoholic hepatitis, current or recent (within 2 months before Day 0) history of significant gastrointestinal disease
18. Clinical evidence of severe ascites, as judged by the Investigator
19. A history of surgical portosystemic shunt
20. For subjects in the healthy control group only:

    * A seated systolic blood pressure (SBP) of < 90 or > 140 mmHg, confirmed by repeat measurement
    * A seated diastolic blood pressure (DBP) of < 40 or > 90 mmHg
    * A history of vitamin preparation or supplement use (including St. John's Wort and ginseng) within 7 days prior to Day 0, or caffeine and methylxanthine (e.g., tea, chocolate) containing foods/beverages within 48 h prior to Day 0
    * A history of prescription or over-the-counter (OTC) drug use within 7 days or 5 half lives of the drug, whichever was longer, prior to Day 0
    * A history of liver disease or liver injury as indicated by an alanine aminotransferase (ALT), aspartate aminotransferase (AST), > 2.5 × the upper limit of normal (ULN) at Screening, or serum bilirubin > 1.5 × ULN
    * Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
21. For subjects in the hepatic impairment group only:

    * A seated SBP of < 80 or > 160 mmHg, confirmed by repeat measurement
    * A seated DBP of < 40 or > 100 mmHg
    * A history of any new prescription medication within 30 days prior to Day 0
    * A history of fluctuating or rapidly deteriorating hepatic function or the production of widely varying or worsening clinical and/or laboratory signs of hepatic impairment within the screening period
22. Any other serious medical condition that, in the opinion of the Investigator, would pose a significant risk to the subject or interfere with the interpretation of safety, PK, or PD data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. P. Lock, M.D., Study Director — Theracos Sub, LLC
Locations (2):
- United States (2):
  - Clinical Research Site 1, Boston, Massachusetts
  - Clinical Research Site 2, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Hepatic Function: Healthy subjects with normal hepatic function. Each subject will receive a single oral dose of bexagliflozin, 20 mg.
- Moderate Hepatic Impairment: Subjects with hepatic impairment conforming to the Child-Pugh class B (total score 7-9). Each subject will receive a single oral dose of bexagliflozin tablet, 20 mg
Period: Overall Study
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (4.16) | 59.9 (4.58) | 58.5 (4.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Child-Pugh Total Score [Mean (Standard Deviation); unit: scores on a scale] — The Child-Pugh classification score was used to determine the severity of hepatic impairment. A patient was rated a score of 1 to 3 for each of the 5 categories: encephalopathy, ascites, bilirubin, albumin and INR. The total score was the sum of the scores for each category with a minimum of 5 and a maximum of 15. A subject would have a mild hepatic impairment with a Child-Pugh score of 5 to 6, a moderate impairment with a score of 7 to 9 and a severe impairment with a score of 10 to 15. A subject with normal hepatic function would have a score of 0 assigned.
  scores on a scale | 0 (0) | 8.3 (0.89) | 4.13 (4.30)
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 2 | 2 | 4
  Former Smoker | 3 | 3 | 6
  Non-Smoker | 3 | 3 | 6
Pack Years of Cigarette Smoking [Mean (Standard Deviation); unit: years] — Population: Number analyzed only include current and former smokers
  years
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 5.2 (5.27) | 13.2 (20.09) | 9.23 (14.47)

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Plasma Concentration)
Description: Whole venous blood samples of 6mL were collected from a peripheral vein prior to dosing and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h after administration of bexagliflozin. The pharmacokinetic parameters were estimated from the bexagliflozin plasma concentration data for each subject by non-compartmental analysis (NCA).
Time Frame: Up to 48 hours
Population: The Pharmacokinetic (PK) population included all subjects without major protocol violations who were dispensed the study drug and provided an observation for at least one primary PK endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
ng/mL
  Total Bexagliflozin | 90.8 (34.0) | 96.5 (37.3)
  Unbound Bexagliflozin | 6.0 (45.5) | 6.6 (46.6)
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; Geometric LS Mean was used as PK parameters for total bexagliflozin by hepatic function group; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Point Estimate = 106.22, 90% CI 2-sided [78.34 to 144.02] — Point Estimate is the estimated ratio of exponentiated mean difference of log-transformed PK parameter from ANOVA. Confidence interval is obtained from ANOVA with hepatic function group as a fixed effect, and the subject as a random effect
Statistical Analysis 2: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; Geometric LS Mean was used as PK parameters for unbound bexagliflozin by hepatic function group; Test type: Equivalence — The acceptance range for bioequivalence is 80.00 - 125.00%; Point Estimate = 110.84, 90% CI 2-sided [75.34 to 163.06] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Tmax (Time of Maximum Observed Plasma Concentration)
Description: as for outcome 1
Time Frame: Up to 48 hours
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
hours
  Total Bexagliflozin | 3.00 [2.00 to 3.05] | 3.00 [2.00 to 3.00]
  Unbound Bexagliflozin | 3.00 [2.00 to 3.05] | 3.00 [2.00 to 3.05]

3. Primary Outcome: T1/2 (Apparent Terminal Elimination Half-life)
Description: as for outcome 1
Time Frame: Up to 48 hours
Population: The adjusted r2 value for the regression for Subject 4551383007 (normal hepatic function group) was less than 0.7. The T1/2 was not estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
hours
  Total Bexagliflozin | 9.4 (40.2) | 9.5 (51.0)
  Unbound Bexagliflozin: number analyzed (Participants) | 7 | 8
  Unbound Bexagliflozin | 11.3 (44.1) | 10.6 (37.7)

4. Primary Outcome: AUC0-inf (Area Under the Plasma Concentration-time Curve From Time 0 to Infinity)
Description: as for outcome 1
Time Frame: Up to 48 hours
Population: The adjusted r2 value for the regression for Subject 4551383007 (normal hepatic function group) was less than 0.7. The AUC0-inf was not estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
ng*h/mL
  Total Bexagliflozin | 695.8 (25.3) | 893.0 (32.2)
  Unbound Bexagliflozin: number analyzed (Participants) | 7 | 8
  Unbound Bexagliflozin | 47.9 (31.0) | 63.3 (38.9)
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; Geometric LS Mean was used as PK parameters for total bexagliflozin by hepatic function group; Test type: Equivalence — The acceptance range for bioequivalence is 80.00 - 125.00%; Point Estimate = 128.34, 90% CI 2-sided [99.98 to 164.73] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; Geometric LS Mean was used as PK parameters for unbound bexagliflozin by hepatic function group; Test type: Equivalence — The acceptance range for bioequivalence is 80.00 - 125.00%; Point Estimate = 132.16, 90% CI 2-sided [96.46 to 181.08] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Urinary Glucose Excretion 0-48 Hours
Description: Pre-dose urine samples were collected from -12 to 0 h for baseline measurement of pharmacodynamic parameters. Post-dose urine samples were collected without preservative in four batches: 0 to 12 h, 12 to 24 h, 24 to 36h, and 36 to 48 h after dosing. Urine aliquots were prepared from well mixed collections for the assessment of pharmacodynamics.
Time Frame: 0-48 hours
Population: The Pharmacodynamic (PD) Population included all subjects without major protocol violations who were dispensed the study drug and produced at least the first 12 h post-dose urine. The PD Population was used to summarize the PD parameters. One subject in the Normal Hepatic Function group did not have the urinary glucose concentration measurement on the 36 to 48-hour urine collection.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
g
  Pre-dose (-12 - 0 hours) | 0.04 (0.045) | 0.91 (2.464)
  0 - 12 hours post-dose | 37.76 (7.253) | 29.57 (8.492)
  12 - 24 hours post-dose | 21.99 (5.780) | 19.25 (6.311)
  24 - 36 hours post-dose | 26.76 (14.588) | 20.96 (11.340)
  36 - 48 hours post-dose: number analyzed (Participants) | 7 | 8
  36 - 48 hours post-dose | 5.87 (4.785) | 5.11 (5.165)
  0 - 24 hours post-dose | 59.75 (12.497) | 48.82 (12.405)
  0 - 48 hours post-dose: number analyzed (Participants) | 7 | 8
  0 - 48 hours post-dose | 91.92 (28.142) | 74.89 (25.410)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from Day 0 up to Day 16 after drug administration
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Hepatic Function (N=8) | Moderate Hepatic Impairment (N=8)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator does not have the right to publish trial results.

DOCUMENTS (2):
  • Study Protocol (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT03557658/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT03557658/SAP_001.pdf